CLINICAL TRIAL: NCT01059760
Title: Expression of Longevity Genes in Response to Extended Fasting
Acronym: FEELGOOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 154-002
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2011-03

CONDITIONS: Cardiovascular Disease
Keywords: Fasting; Short-term starvation; Diet; Coronary artery disease
MeSH Terms: conditions — Cardiovascular Diseases; Fasting; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fasting Day First (Other): 28±4 hours of water-only fasting followed by 28±4 hours fed
  Interventions: Behavioral: Fasting First
- Fed Day First (Other): 28± 4 hours fed followed by 28± 4 hours of fasting
  Interventions: Behavioral: Fed First

INTERVENTIONS:
Behavioral: Fasting First — 28±4 hours of water-only fasting followed by 28±4 hours fed
  Arms: Fasting Day First
Behavioral: Fed First — 28± 4 hours fed followed by 28± 4 hours of fasting
  Arms: Fed Day First

SUMMARY:
The purpose of this study is to evaluate the effect of fasting on physical changes associated with cardiovascular disease.

DETAILED DESCRIPTION:
Coronary heart disease (CHD) is the largest contributor to morbidity and mortality in the Western world and is associated with high-calorie diet, high body mass, and a variety of other factors. CHD can lead to myocardial infarction (MI) and other embolic events. A growing body of evidence suggests that relatively low caloric intake in the diets of a variety of animals increases longevity and preliminary evidence among humans indicates that such caloric restriction reduces risk factors for CHD, including cholesterol levels, blood pressure, glucose, and obesity. Caloric restriction has also been shown to alter the expression of certain genes, especially the forkhead box (FOX) O and sirtuin (SIRT) genes whose over-expression has been shown to increase longevity in animal models. Extended avoidance of caloric intake, also called fasting or short-term starvation, has been shown to increase expression of the FOXA genes that have similar sequence and function as the FOXO genes and that have been shown to increase longevity among animals regardless of FOXO function. We recently demonstrated that the risk of CHD was significantly lower among patients who reported a history of routine periodic extended fasting. The two primary hypotheses for this observation are that fasting may improve individual ability to control dietary intake or that fasting may initiate a cascade of protective mechanisms that preserve cellular and metabolic health.

ELIGIBILITY:
Inclusion Criteria:

1. The volunteer (male or non-pregnant female, any ethnicity) must be >18 years of age.
2. The volunteer must either have a body mass index of 25.0-35.0 kg/m2 or the combination of a body mass index of 18.5-24.9 kg/m2 and two or more previously or currently measured symptoms of the metabolic syndrome (fasting glucose≥110 mg/dL, triglycerides≥150 mg/dL, high-density lipoprotein cholesterol<40 mg/dL in males or <50 mg/dL in females, systolic blood pressure≥130 mmHg or diastolic blood pressure≥85 mmHg, or waist circumference≥40 inches in males or ≥36 inches in females [glucose and cholesterol levels may be self-reported]).
3. The volunteer has not routinely participated in caloric restriction (deliberate limitation of caloric intake of <80% than the FDA-recommended daily caloric intake) within the last 2 years, has not participated in extended fasting (>12 hours at a time) for at least a year, and does not deliberately skip meals as a routine dietary practice.

Exclusion Criteria:

1. Body mass index <18.5 or >35 kg/m2.
2. Current active cancer treatment, treatment with immunosuppressive medications, or solid organ transplantation within 1 year.
3. Presence of immunosuppressive disease, myocardial infarction, peripheral vascular disease, or stroke within the past year.
4. Use of insulin.
5. Although it is unlikely fasting will harm the pregnant or lactating woman, the dietary restrictions placed on the participant for the duration of the study may conflict with dietary recommendations for pregnant or lactating women. Women of child bearing potential, therefore, will meet an exclusion if they become pregnant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Horne, PhD, Principal Investigator — Intermountain Medical Center
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

REFERENCES:
- [Background] Horne BD, May HT, Anderson JL, Kfoury AG, Bailey BM, McClure BS, Renlund DG, Lappe DL, Carlquist JF, Fisher PW, Pearson RR, Bair TL, Adams TD, Muhlestein JB; Intermountain Heart Collaborative Study. Usefulness of routine periodic fasting to lower risk of coronary artery disease in patients undergoing coronary angiography. Am J Cardiol. 2008 Oct 1;102(7):814-819. doi: 10.1016/j.amjcard.2008.05.021. Epub 2008 Jul 10. PMID 18805103
- [Derived] Horne BD, Anderson JL, May HT, Bair TL, Le VT, Iverson L, Knowlton KU, Muhlestein JB. Weight loss-independent changes in human growth hormone during water-only fasting: a secondary evaluation of a randomized controlled trial. Front Endocrinol (Lausanne). 2025 Feb 7;15:1401780. doi: 10.3389/fendo.2024.1401780. eCollection 2024. PMID 39991046
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717
- [Derived] Horne BD, Muhlestein JB, Lappe DL, May HT, Carlquist JF, Galenko O, Brunisholz KD, Anderson JL. Randomized cross-over trial of short-term water-only fasting: metabolic and cardiovascular consequences. Nutr Metab Cardiovasc Dis. 2013 Nov;23(11):1050-7. doi: 10.1016/j.numecd.2012.09.007. Epub 2012 Dec 7. PMID 23220077

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fasting Day First | Fed Day First
Started | 16 | 14
Completed | 16 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fasting Day First | Fed Day First | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (13.6) | 44.0 (14.0) | 43.6 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.4 (7.1) | 27.3 (6.1) | 27.8 (1.3)
Hemoglobin A1C [Mean (Standard Deviation); unit: percentage] | 5.5 (0.3) | 5.3 (0.3) | 5.4 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Participant Glucose When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
mg/dL | 83.3 (15.8) | -8.0 (15.4) | 5.9 (16.6)

2. Primary Outcome: Change From Baseline in Participant Human Growth Hormone (HGH) When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
ng/mL | 0.32 (0.47) | 1.54 (2.63) | -1.14 (1.66)

3. Primary Outcome: Change From Baseline in Participant Insulin When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: mU/L
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
mU/L | 23.6 (17.8) | -19.0 (29.3) | -1.6 (16.2)

4. Primary Outcome: Change From Baseline in Participant Homeostasis Model Assessment-Insulin Resistance (HOMA-IR) When Fasting and Fed
Description: HOMA-IR is used to measure the severity of insulin resistance. Healthy Range: 1.0 (0.5-1.4) Less than 1.0 is optimal Above 1.9 indicates early insulin resistance Above 2.9 indicates significant insulin resistance
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
units on a scale | 0.66 (0.051) | -0.35 (0.53) | -.02 (0.30)

5. Primary Outcome: Change From Baseline in Participant Glycogen-Like Protein-1 (GLP-1) When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
ng/mL | 1.77 (0.79) | -0.27 (0.51) | 0.07 (0.51)

6. Primary Outcome: Change From Baseline in Participant Adiponectin When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: ratio of high molecular to total
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
ratio of high molecular to total | 0.34 (0.17) | 0.02 (0.25) | -0.07 (0.25)

7. Primary Outcome: Change From Baseline in Participant Fibroblast Growth Factor-21 (FGF-21) When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
pg/mL | 190.3 (261.4) | -41.7 (128.9) | 9.5 (108.8)

8. Primary Outcome: Change From Baseline in Participant White Blood Cell Count (WBC) When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: cells/mL
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
cells/mL | 6.0 (1.4) | 0.32 (1.31) | -0.12 (1.48)

9. Primary Outcome: Change From Baseline in Participant Hemoglobin When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
g/dL | 14.3 (1.3) | 0.46 (0.37) | -0.39 (0.52)

10. Primary Outcome: Change From Baseline in Participant Red Blood Cell Count (RBC) When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: cells x 10^6/mL
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
cells x 10^6/mL | 4.7 (0.4) | 0.15 (0.13) | -0.11 (0.17)

11. Primary Outcome: Change From Baseline in Participant Hematocrit When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: % of red blood cells to whole blood
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
% of red blood cells to whole blood | 41.6 (3.6) | 1.3 (1.3) | -1.1 (1.5)

12. Primary Outcome: Change From Baseline in Participant Platelet Count When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: cells x 10^3/mL
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
cells x 10^3/mL | 253.5 (58.2) | 2.8 (16.3) | 0.9 (13.8)

13. Primary Outcome: Change From Baseline in Participant Mean Corpuscular Volume (MCV) When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
fL | 89.11 (3.56) | -0.12 (0.68) | -0.18 (0.73)

14. Primary Outcome: Change From Baseline in Participant Mean Corpuscular Hemoglobin (MCH) When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
pg | 30.66 (1.48) | -0.01 (0.33) | -0.07 (0.40)

15. Primary Outcome: Change From Baseline in Participant Mean Corpuscular Hemoglobin Concentration (MCHC) When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
g/dL | 34.4 (0.5) | 0.02 (0.49) | -0.01 (0.52)

16. Primary Outcome: Change From Baseline in Participant Red Cell Distribution Width (RDW) When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: % of SD of MCV to mean MCV
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
% of SD of MCV to mean MCV | 13.6 (0.82) | -0.04 (0.32) | -0.03 (0.37)

17. Primary Outcome: Change From Baseline in Participant Mean Platelet Volume (MPV) When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
fL | 8.17 (0.83) | 0.02 (0.49) | 0.03 (0.26)

18. Primary Outcome: Change From Baseline in Participant Bicarbonate When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
mmol/L | 27.0 (2.5) | -1.4 (1.7) | 0.9 (2.2)

19. Primary Outcome: Change From Baseline in Participant Sodium When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
mmol/L | 139.1 (2.0) | -1.4 (2.1) | 0.7 (2.0)

20. Primary Outcome: Change From Baseline in Participant Chloride When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
mmol/L | 103.7 (2.7) | -1.3 (2.0) | 0.9 (2.3)

21. Primary Outcome: Change From Baseline in Participant Blood Urea Nitrogen (BUN) When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
mg/dL | 16.0 (3.7) | -1.2 (3.9) | 1.8 (2.6)

22. Primary Outcome: Change From Baseline in Participant Calcium When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
mg/dL | 9.4 (0.3) | 0.18 (0.34) | -0.12 (0.33)

23. Primary Outcome: Change From Baseline in Participant Potassium When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
mmol/L | 4.29 (0.28) | -0.02 (0.30) | 0.02 (0.32)

24. Primary Outcome: Change From Baseline in Participant Creatinine When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
mg/dL | 0.848 (0.118) | 0.005 (0.09) | 0.002 (0.06)

25. Primary Outcome: Change From Baseline in Participant Total Cholesterol (TC) When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
mg/dL | 190.7 (30.7) | 9.5 (10.6) | -4.8 (11.0)

26. Primary Outcome: Change From Baseline in Participant Low-Density Lipoprotein Cholesterol (LDL-C) When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
mg/dL | 103.8 (33.8) | 23.1 (35.1) | -10.3 (28.2)

27. Primary Outcome: Change From Baseline in Participant High-Density Lipoprotein Cholesterol (HDL-C) When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
mg/dL | 55.9 (14.3) | 3.7 (5.3) | -1.0 (3.6)

28. Primary Outcome: Change From Baseline in Participant Triglycerides When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
mg/dL | 134.2 (77.0) | -52.4 (55.5) | 11.2 (38.1)

29. Primary Outcome: Change From Baseline in Participant TC/HDL Ratio When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
ratio | 3.63 (1.15) | -3.3 (17.7) | 0.0 (0.2)

30. Primary Outcome: Change From Baseline in Participant Weight When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
kg | 81.3 (25.0) | -1.5 (0.9) | 0.5 (0.9)

31. Primary Outcome: Change From Baseline in Participant Waist Circumference When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
cm | 86.7 (16.7) | -0.57 (1.4) | 0.54 (3.0)

32. Primary Outcome: Change From Baseline in Participant Systolic Blood Pressure (SBP), Supine When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
mmHg | 114.0 (13.6) | -3.1 (8.4) | 1.0 (9.6)

33. Primary Outcome: Change From Baseline in Participant Diastolic Blood Pressure (DBP), Supine When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
mmHg | 67.2 (8.8) | 1.7 (7.4) | -1.2 (8.9)

34. Primary Outcome: Change From Baseline in Participant High Sensitivity C-Reactive Protein (hsCRP) When Fasting and Fed
Time Frame: Baseline and 3 days
Measure: Median (Standard Error); unit: mg/L
Arm/Group | Baseline Value | Change While Fasting | Change When Fed
Number analyzed (Participants) | 30 | 30 | 30
mg/L | 1.35 (0.96) | 0.00 (0.44) | -0.10 (0.24)

ADVERSE EVENTS:
Time Frame: 3 days
Groups:
- Fasting Day First: Includes those who fasted on the 1st day.
- Fed Day First: Includes those who fasted on the 2nd day.
Arm/Group | Fasting Day First | Fed Day First
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 2/16 | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fasting Day First (N=16) | Fed Day First (N=14)
Mild Headache (General disorders) | 1 (1) | 1 (1)
Migraine (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes